CLINICAL TRIAL: NCT07128927
Title: Assessing the Feasibility of Web-based Insomnia Treatment Among Prostate Cancer Survivors
Acronym: SIESTA-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007350
Record Dates: First submitted 2025-08-05; First posted 2025-08-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Insomnia
Keywords: insomnia; Sleep Healthy Using the Internet (SHUTi); prostate cancer survivorship; cognitive behavioral therapy for insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Healthy Using the Internet (SHUTi) (Experimental): SHUTi provides 6 sessions of 45-60 minutes in length delivered over the course of 6-9 weeks. The program tailors recommendations based on sleep diary data provided by each participant.
  Interventions: Behavioral: Sleep Healthy Using the Internet (SHUTi)
- Patient education (Placebo Comparator): Static information about insomnia provided on a patient education website
  Interventions: Behavioral: Patient education

INTERVENTIONS:
Behavioral: Sleep Healthy Using the Internet (SHUTi) — Web-based, self-administered, and interactive cognitive behavioral therapy for insomnia
  Other Names: Cognitive behavioral therapy for insomnia; CBT-i
  Arms: Sleep Healthy Using the Internet (SHUTi)
Behavioral: Patient education — Website that describes insomnia, including factors that may increase or decrease insomnia symptoms, and provides information about addressing insomnia symptoms.
  Other Names: Sleep hygiene
  Arms: Patient education

SUMMARY:
This pilot study will recruit Black/African American prostate cancer survivors into a clinical trial and will randomize each person to 1 of 2 possible treatments - an internet-based treatment for insomnia called Sleep Healthy Using the Internet (SHUTi) or an educational website. SHUTi provides the treatment - cognitive behavioral therapy for insomnia - across 6 lessons, while the educational website is like an online patient brochure. The study will examine the feasibility of SHUTi to improve sleep and well-being among Black prostate cancer survivors. It will also examine whether SHUTi is acceptable to these survivors and will compare the effect of SHUTi versus the educational website on insomnia and non-insomnia patient-reported outcomes.

DETAILED DESCRIPTION:
Insomnia is a risk factor for poor physical, cognitive, and psychosocial outcomes, including depression, anxiety, frailty, and diminished cognitive function, especially among cancer survivors. Although Cancer treatment, including androgen deprivation therapy, may increase insomnia symptoms and the prevalence of insomnia among prostate cancer survivors is estimated to be 25-39%. Prostate cancer has the highest incidence rate and second highest mortality rate among men in the U.S. with a highest burden of both incidence and mortality among Black men compared to men of other racial/ethnic groups. However, few studies have examined treatment of insomnia in this population. Insomnia is associated with greater symptom burden (i.e., multiple concurrent symptoms, such as depression, anxiety, fatigue, pain, cognition) among prostate cancer survivors, so treating insomnia may provide an opportunity to improve well-being in this population.

Cognitive Behavioral Therapy for Insomnia (CBT-I) has demonstrated substantial and persistent improvements in insomnia severity among cancer survivors such that the National Comprehensive Cancer Network (NCCN) recommends it "as the preferred treatment for insomnia." Trials to develop and test web-based and digital CBT-I interventions have shown non-inferiority to in-person administration by a trained therapist and increase availability of insomnia treatment to more patients. Recent NCCN guidelines note that improving sleep may provide additional benefits by resulting in less fatigue, better mood, better quality of life, and improved survival. However, to date, this accessible and interactive intervention has not been investigated among prostate cancer survivors.

This study uses the Sleep Healthy Using the Internet (SHUTi) program to provide CBT-I via the internet. SHUTi is self-administered and interactive with 6 weekly 45-60 minute sessions delivered over the course of 9 weeks. The program uses sleep diary data provided by each participant to tailor recommendations. Prostate cancer survivors participating in this pilot study will be randomized to receive access to SHUTi or to a patient education website. All participants will complete study visits and data collection, including sleep diaries and questionnaires, at baseline and post-intervention (10-12 weeks later).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* Self-identifies as Black/African American
* Diagnosed with invasive prostate cancer (AJCC stages I-IV) within 5 years
* Has not received surgery, chemotherapy, or radiation within the previous 3 months
* Has a smart phone, tablet, or computer with reliable internet access or willing to attend a weekly study appointment and to complete a weekly phone call
* Has clinically relevant insomnia symptoms (i.e., score ≥10 on the Insomnia Severity Index)
* Able to read and understand English

Exclusion Criteria:

* Employed in an occupation where sleep restriction could be a harm to themselves or others
* Actively employed in shift work
* Diagnosed with a severe/major psychiatric disorder
* Diagnosed with a seizure disorder or recently (≤12 months) experienced a seizure
* Unable to consent

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study protocol | 10-12 weeks
  Assessed via:
  * the percentage of survivors screened as eligible who consent to participate,
  * the percentage of actual vs. planned participants enrolled, and
  * the percentage of enrolled participants complete follow-up data collection
Acceptability of intervention | 10-12 weeks
  Assessed via the theoretical framework of acceptability questionnaire (range: 5-35, higher score = greater acceptability)

SECONDARY OUTCOMES:
Efficacy of intervention | 10-12 weeks
  Assessed via change in the Insomnia Severity Index score (range: 0-28, higher score = more insomnia symptoms) from baseline to post-intervention

OTHER OUTCOMES:
Impact on non-insomnia patient-reported outcomes | 10-12 weeks
  Assessed via change in total number of reported non-insomnia patient-reported symptoms from baseline to post-intervention (range: 0-5, higher number = greater change in symptoms):
  * Functional Assessment of Cancer Therapy - Prostate (range: 0-156, higher score = better quality of life, score below baseline median = 1 PRO)
  * Male Depression Risk Scale short form (range: 0-154, higher score = greater symptoms of depression, score above baseline median = 1 PRO)
  * 18-item Memorial Anxiety Scale for Prostate Cancer (range: 0-54, higher score = greater anxiety symptoms, score above baseline median = 1 PRO)
  * Functional Assessment of Cancer Therapy - Cognitive Function - Perceived Cognitive Impairments (range: 0-72, higher score = better cognitive function, score below baseline median = 1 PRO)
  * Hot Flash Related Daily Interference Scale (range: 0-100, higher score = more interference, score above baseline median = 1 PRO)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Bai P. Application and Mechanisms of Internet-Based Cognitive Behavioral Therapy (iCBT) in Improving Psychological State in Cancer Patients. J Cancer. 2023 Jul 3;14(11):1981-2000. doi: 10.7150/jca.82632. eCollection 2023. PMID 37497400
- [Background] Gonzalez BD, Small BJ, Cases MG, Williams NL, Fishman MN, Jacobsen PB, Jim HSL. Sleep disturbance in men receiving androgen deprivation therapy for prostate cancer: The role of hot flashes and nocturia. Cancer. 2018 Feb 1;124(3):499-506. doi: 10.1002/cncr.31024. Epub 2017 Oct 26. PMID 29072790
- [Background] Leger P, Frencher S Jr, Nauseef JT, Jones B, Bilen MA, Brown A Jr, Ullah A, McDevitt S, Tsao CK. A multi-perspective study assessing Black and African American participation barriers in prostate cancer clinical trials. Future Oncol. 2025 Apr;21(8):967-973. doi: 10.1080/14796694.2025.2467519. Epub 2025 Feb 24. PMID 39992723
- [Background] Ritterband LM, Thorndike FP, Gonder-Frederick LA, Magee JC, Bailey ET, Saylor DK, Morin CM. Efficacy of an Internet-based behavioral intervention for adults with insomnia. Arch Gen Psychiatry. 2009 Jul;66(7):692-8. doi: 10.1001/archgenpsychiatry.2009.66. PMID 19581560

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT07128927/Prot_SAP_000.pdf